CLINICAL TRIAL: NCT06362642
Title: A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effect of Coadministration of Itraconazole on the Pharmacokinetics of PC14586 in Healthy Participants
Brief Title: A Study to Investigate the Effects of Itraconazole on the Pharmacokinetics of PC14586 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PMV Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PMV-586-105
Record Dates: First submitted 2024-03-25; First posted 2024-04-12 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Y220C; PC14586; PMV Pharma; PMV; itraconazole; rezatapopt; Phase 1; CYP3A4
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: The treatments will be: Day 1: single oral dose of PC14586, Day 20: oral dose of itraconazole BID, Day 21-22: single oral dose of itraconazole QD, Day 23: single oral dose of PC14586 and single oral dose of itraconazole, Day 24-27: single oral dose of itraconazole QD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PC14586 and Itraconazole (Experimental): Healthy participants will receive a single, oral dose of PC14586 on day 1. On day 20, participants will receive BID oral doses of itraconazole. On days 21-22, participants will receive a single, oral dose of itraconazole. On day 23, participants will receive a single, oral dose of PC14586 and a single oral dose of itraconazole. On days 24-27, participants will receive a single, oral dose of itraconazole.
  Interventions: Drug: PC14586; Drug: Itraconazole

INTERVENTIONS:
Drug: PC14586 — First-in-class, oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation.
  Other Names: rezatapopt
Drug: Itraconazole — Antifungal treatment that is a potent inhibitor of CYP3A4.

SUMMARY:
The purpose of this study is to assess the effect of PC14586 pharmacokinetics when co administered with itraconazole in healthy participants.

DETAILED DESCRIPTION:
PC14586 is a first-in-class, oral, small molecule p53 reactivator that is selective for the TP53 Y220C mutation.

This is a Phase 1, open-label, fixed-sequence study to investigate the effect of coadministration of itraconazole on the pharmacokinetics (PK) of PC14586 (rezatapopt) in healthy male and female participants. Potential participants will be screened to assess their eligibility to enter the study within 56 days prior to the first dose administration. Participants will be admitted into the study site on Day -1 and be confined to the study site until discharge on Day 33. Participants will return to the study site for PK sample collection on Day 37 and a follow-up visit and PK sample collection on Day 42.

Approximately 16 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking males and females, aged 18-55 years of age, with BMI between 18.0 and 32.0 kg/m2 inclusive.
2. In good health, determined by no clinically significant findings from medical history and evaluations at screening and check-in as assessed by the investigator.
3. Females of non-childbearing potential, males who agree to a highly effective method of contraception from first dose through 3 months after end of study visit.
4. Participants who are able to swallow tablets and capsules.
5. Participants who are capable and willing of giving signed informed consent.

Exclusion Criteria:

1. Participants with significant medical history or clinical manifestation of any medical condition, disease or disorder, as determined by the investigator.
2. History of significant hypersensitivity, intolerance, or allergy to itraconazole or any of the excipients or to medicinal products with similar chemical structures, food or other substance.
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
4. Participant has blood pressure >140 mmHg systolic or >90 mmHg diastolic at screening or Day -1.
5. Prolonged QT interval corrected for heart rate using Fridericia's correction >450 ms for males and >470 ms for females at screening.
6. Positive hepatitis panel and/or positive human immunodeficiency virus test.
7. Abnormalities in liver function test ALT or AST >1.5 × upper limit of normal.
8. Administration of any vaccine including coronavirus disease 2019 vaccine in the past 14 days prior to check-in.
9. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to check-in.
10. Use or intend to use any prescription medications/products or any nonprescription medications/products within 14 days prior to check-in.
11. Participation in a clinical study involving last administration of an investigational drug (new chemical entity) in the past 30 days prior to dosing, or within 5 half-lives of the IMP, whichever is longer, or have previously received PC14586.
12. Participant has a history of alcohol or drug/chemical abuse within 2 years prior to check-in and/or is unwilling to avoid use of caffeine or alcohol or caffeine-containing foods or alcohol-containing foods, medications, or beverages, within 48 hours prior to check-in until the follow up visit.
13. Use of tobacco- or nicotine-containing products (cigarettes, snuff, chewing tobacco, cigars, pipes, vaporizer, or nicotine-replacement products such as nicotine chewing gum and nicotine patches) within 3 months prior to check-in, or positive cotinine at screening or check-in.
14. Participants with a germline TP53 Y220C mutation at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
Characterize the Maximum Plasma Concentration (Cmax) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the Cmax of PC14586 when co-administered with itraconazole in plasma.
Characterize the total drug exposure (AUC0-inf) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-inf of PC14586 when co-administered with itraconazole in plasma.
Characterize the time to peak drug concentration (Tmax) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the Tmax of PC14586 when co-administered with itraconazole in plasma.
Characterize the total drug exposure from time zero to 24 hours (AUC0-24) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-24 of PC14586 when co-administered with itraconazole in plasma.
Characterize the total drug exposure from time zero to the last timepoint (AUC0-t) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-t of PC14586 when co-administered with itraconazole in plasma.
Characterize the half-life (t1/2) of PC14586 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the t1/2 of PC14586 when co-administered with itraconazole in plasma.

SECONDARY OUTCOMES:
Characterize the Maximum Plasma Concentration (Cmax) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the Cmax of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Characterize the total drug exposure (AUC0-inf) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-inf of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Characterize the time to peak drug concentration (Tmax) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the Tmax of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Characterize the total drug exposure from time zero to 24 hours (AUC0-24) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-24 of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Characterize the total drug exposure from time zero to the last timepoint (AUC0-t) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the AUC0-t of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Characterize the half-life (t1/2) of PC14586 metabolites M13 and M14 when co-administered with itraconazole in healthy participants. | 6 weeks
  Determine the t1/2 of PC14586 metabolites M13 and M14 when co-administered with itraconazole in plasma.
Identification of the incidence of treatment emergent adverse events (TEAE) of PC14586 when administered alone and co-administered with itraconazole in healthy participants. | 6 weeks
  Identify the incidence of TEAEs of PC14586 alone or when co-administered with itraconazole.
Identification of vital sign abnormalities after administration of PC14586 alone and when co-administered with itraconazole in healthy participants. | 6 weeks
  Identify the number of participants with abnormal vital signs.
Identification of 12-lead electrocardiogram (ECG) abnormalities after administration of PC14586 alone and when co-administered with itraconazole in healthy participants. | 6 weeks
  Identify the number of participants with abnormal ECG results.
Identification of laboratory abnormalities based on hematology and clinical chemistry after administration of PC14586 alone and when co-administered with itraconazole in healthy participants. | 6 weeks
  Identify the number of participants with an incidence of laboratory abnormalities in test results.

CONTACTS AND LOCATIONS:
Locations (1):
- Fortrea, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No